CLINICAL TRIAL: NCT01101997
Title: Non-Invasive Reduction of Abdominal Fat Utilizing the JUNO Applicator
Brief Title: Non-Invasive Reduction of Abdominal Fat
Acronym: JUNO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeltiq Aesthetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ZA10-001
Record Dates: First submitted 2010-04-05; First posted 2010-04-12 (Estimated); Results first posted 2020-12-21 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-08

CONDITIONS: Fat Reduction
Keywords: Lipolysis; Cryolipolysis; Fat Reduction
MeSH Terms: interventions — Lipectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Experimental: Abdomen Treatment Group (Experimental): All subjects were treated on the abdomen with the CoolSculpting system.
  Interventions: Device: The Zeltiq System

INTERVENTIONS:
Device: The Zeltiq System — Noninvasive cooling is applied to the treatment area with a defined cooling rate and duration.
  Other Names: Cryolipolysis; Lipolysis

SUMMARY:
This study is being performed to reduce unwanted abdominal fat using a new applicator for the Zeltiq System.

DETAILED DESCRIPTION:
The primary objective of the study is to achieve a discernable change to the contour of the abdominal area treated with the JUNO applicator that is consistent with that documented during a clinical study of a previous applicator used to treat lovehandles.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects > 18 years of age.
2. Subject has clearly visible fat on the abdomen.
3. Subject has not had weight change exceeding 10 pounds in the preceding month.
4. Subject agrees to maintain their weight (i.e., within 5 pounds) by not making any major changes in their diet or lifestyle during the course of the study.
5. Subject has read and signed a written informed consent form.

Exclusion Criteria:

1. Subject has had a surgical procedure(s) in the area of intended treatment in the past 6 months.
2. Subject has had an invasive fat reduction procedure (e.g., liposuction, abdominoplasty, mesotherapy) in the area of intended treatment within the past year.
3. Subject has had a non-invasive fat reduction procedure in the area of intended treatment within the past 6 months.
4. Subject has a known history of subcutaneous injections into the area of intended treatment (e.g., heparin, insulin) within the past month.
5. Subject has a known history of cryoglobulinemia, cold urticaria, or paroxysmal cold hemoglobinuria.
6. Subject has a known history of Reynaud's disease, or any known condition with a response to cold exposure that limits blood flow to the skin.
7. Subject has a history of bleeding disorder or is taking any medication that in the investigator's opinion may increase the subject's risk of bruising.
8. Subject body mass index (BMI) exceeds 40. BMI is defined as weight in pounds multiplied by 703 divided by the square of the height in inches.
9. Subject is taking or has taken diet pills or supplements within the past month.
10. Subject has any dermatological conditions or scars in the location of the treatment sites that may interfere with the treatment or evaluation.
11. Subject is pregnant or intending to become pregnant in the next 6 months.
12. Subject is lactating or has been lactating in the past 6 months.
13. Subject is unable or unwilling to comply with the study requirements.
14. Subject is currently enrolled in a clinical study of any other unapproved investigational drug or device.
15. Any other condition or laboratory value that would, in the professional opinion of the investigator, potentially affect the subject's response or the integrity of the data or would pose an unacceptable risk to the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-03-30 (Actual); Primary Completion 2010-09-28 (Actual); Study Completion 2010-12-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Laser and Skin Surgery of Northern California, Sacramento, California
  - Flor Mayoral, M.D., Coral Gables, Florida
  - Maryland Laser, Skin and Vein Institute, Hunt Valley, Maryland
  - Skin Care Physicians of Chestnut Hill, Chestnut Hill, Massachusetts
  - Zel Skin and Laser Specialist LLC, Edina, Minnesota

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Zeltiq System Treatment Group: The treatment group consists of all subjects treated with the Zeltiq System for the reduction of abdominal fat.
Period: Overall Study
Arm/Group | Zeltiq System Treatment Group
Started | 60
Completed | 58
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: The baseline analysis population included all subjects enrolled in the study.
Arm/Group | Zeltiq System Treatment Group
Number analyzed (Participants) | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 60
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.0 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 60
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — The Fitzpatrick Skin Type scale is a numerical classification schema for human skin color, developed as a way to estimate the response of different skin types of skin to ultraviolet (UV) light. Fitzpatrick skin type characteristics are present at birth. The scale is composed of six skin type classifications for FST I to FST VI.
  There is no additional value in the skin type scale, e.g., a FST VI classification is no more or less valuable than a classification of FST I, FST II, FST III, FST IV or FST V.
  Participants
    FST I-Always burns, never tans | 5
    FST II- Burns easily, tans poorlyy | 22
    FST III- Tans after initially burning | 21
    FST IV- Burns minimally, tans easily | 10
    FST V- Rarely burns, tans darkly easily | 1
    FST VI- Never burns | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Pre-treatment Images Correctly Identified
Description: Change in the treated vs. untreated areas will be assessed by observation of changes in surface contour and/or fat volume by an independent photo review of pre-treatment and post-treatment images of the treated areas. Reviewers will be practicing dermatologists or plastic surgeons. All reviewers will be blinded to post-treatment vs. baseline untreated area. The order in which images will be presented will be randomized; for each subject placement of the baseline, pre-treatment image will be randomized for each pair of subject images. Reviewers will be asked to select the baseline photos for each subject photo series and record selections on a data collection form. The expected success rate is an average 80% correct identification by the three reviewers.
Time Frame: 16 weeks
Population: The per protocol population are those subjects who were treated with the Zeltiq CoolSculping System and maintained weight as specified in the protocol.
Measure: Count of Units; unit: photos
Units Other Than Participants: photos
Groups:
- Zeltiq System Treatment Group: The per protocol population consists of all evaluable subjects treated with the Zeltiq System for the reduction of abdominal fat and whose weight change was within 5 pounds of baseline weight.
Arm/Group | Zeltiq System Treatment Group
Number analyzed (Participants) | 50
Number analyzed (photos) | 150
photos | 128
Statistical Analysis 1: Comparison: Zeltiq System Treatment Group; H0: p= 0.6 and Ha: p ≠ 0.6; Test type: Superiority; p < 0.001, Chi-squared; sucess proportion = .853, 95% CI 2-sided [.773 to .910]

2. Secondary Outcome: Change in the Fat Layer of the Treated Area as Measured by Ultrasound
Description: Change in the fat layer thickness will be calculated by comparison of pre-treatment and 16 week post-treatment ultrasound measurements taken in the area treated with the device, and in the adjacent untreated control area. The Sponsor's standardized techniques for obtaining ultrasound imaging will be used. Overall fat layer thickness changes were normalized for each subject by subtracting the change in control from the change in treated area to remove the influence of weight variations. Results indicate the fat layer reduction in mm.
Time Frame: 16 weeks
Population: All subjects who completed treatment with the Zeltiq System, independent of weight changes, were included in the analysis population.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Experimental: Abdomen Treatment Group
Number analyzed (Participants) | 58
mm | -1.9 (2.49)
Statistical Analysis 1: Comparison: Experimental: Abdomen Treatment Group; Test type: Other; Mean Difference (Net) = -1.9, Standard Deviation 2.49

3. Secondary Outcome: Subject Satisfaction
Description: Subject satisfaction with the Zeltiq procedure as determined by the results of a subjects satisfaction questionnaire at the 16 week follow up visit.
Time Frame: 16 weeks
Population: All evaluable subjects that completed the satisfaction questionnaire were included in the analysis.
Measure: Number; unit: percent of positive responses
Arm/Group | Zeltiq System Treatment Group
Number analyzed (Participants) | 58
percent of positive responses
  Procedure somewhat uncomfortable to very comfortab | 88
  Visible change in contour of treated region | 60
  At least a slight difference in fit of clothes | 79
  Overall effect was about, or more than expected | 50
  Overall satisfaction with the procedure | 62
  Would repeat the procedure | 62
  Would have the procedure on different body part | 65
  Would recommend the procedure | 67

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time of enrollment through the 16 week follow-up visit.
Arm/Group | Zeltiq System Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 10/60
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zeltiq System Treatment Group (N=60)
Nausea (Gastrointestinal disorders) | 2 (2)
Pain (General disorders) | 2 (2)
Numbness (Skin and subcutaneous tissue disorders) | 2 (2)
Anxiety (General disorders) | 1 (1)
Vasovagal event (General disorders) | 1 (1)
Headache (General disorders) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No